CLINICAL TRIAL: NCT06584552
Title: Lactobacillus Paracasei LPB27 On Early Childhood Eczema
Brief Title: LaCE (Lactobacillus Paracasei LPB27 On Early Childhood Eczema)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Evolution Health Pty Ltd (Unknown)
Responsible Party: Principal Investigator, Keith Chee Y. Ooi, Professor, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024001_LaCE
Record Dates: First submitted 2024-08-21; First posted 2024-09-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-09

CONDITIONS: Eczema; Allergy
Keywords: Immunology; Microbiome; Paediatrics
MeSH Terms: conditions — Eczema; Hypersensitivity | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactobacillus Paracasei LPB27 (Experimental): Formulation: Lactobacillus paracasei LPB27 (10 billion cfu/ serve) and Maltodextrin (up to 1g).
  Dosage: 1mg daily for 12 weeks. Delivered orally through through breast milk, formula or solid food.
  Interventions: Dietary Supplement: Lactobacillus Paracasei LPB27
- Maltodextrin (Placebo Comparator): Formulation: Maltodextrin 1g
  Dosage: 1mg daily for 12 weeks. Delivered orally through through breast milk, formula or solid food.
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Lactobacillus Paracasei LPB27 — Probiotic
  Arms: Lactobacillus Paracasei LPB27
Other: Maltodextrin — Placebo
  Arms: Maltodextrin

SUMMARY:
The LaCE study is a double-blind, randomised, placebo-controlled trial examining the effectiveness of the probiotic Lactobacillus paracasei LPB27 in treating eczema in young children.

DETAILED DESCRIPTION:
Childhood eczema is a common and chronic, relapsing disease of the skin which affects up to 20% of the paediatric population. Eczema has significant impact on the quality of life of those affected. Its main symptoms are dry skin and intense itching.

There is currently no cure for eczema but there are treatments that try to relieve symptoms. These commonly include topical moisturisers and topical corticosteroids.

Although topical corticosteroids are effective in minimising symptoms, there is a prevailing and universal fear of using topical corticosteroids which is one of the main reasons for poor treatment compliance.

There have been emerging interests in prevention and treatment of eczema through modulation of the gut microbiome. The gut microbiome is a key regulator for the immune system and there is evidence that the composition of gut microbiome may reduce allergies by driving maturation of the immune system. It was shown that people with eczema have different bacteria in their gut compared to people without eczema. Therefore, this study's hypothesis is that administration of oral probiotics will benefit young children with eczema by improving their gut microbiome and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3 months to 3 years old
* Diagnosis: Eczema (atopic dermatitis) diagnosed clinically by a paediatric dermatologist or immunologist.
* Severity: Investigator Global Assessment for Atopic Dermatitis (IGA) severity of 1-3 (almost clear, mild, moderate) and a SCORAD score greater than 8.7.
* Willingness and ability of the subject to comply with the protocol requirements.

Exclusion Criteria:

* Patients on systemic immunosuppression and/or biologic agents (participants who start systemic immunosuppression and/or biologic agents mid-way through the study will be considered to have not achieved treatment success and will be withdrawn, regardless of their SCORAD index scores).
* Mothers who are breastfeeding and on probiotics but not willing to stop probiotics.
* Child already on probiotics and parents not willing to stop during the entire study period (washout period of 4 weeks; including formulas that contains probiotics).
* Eczema complicated by active skin infection e.g. impetigo/cellulitis/ eczema herpeticum (can be considered once active infection resolved).
* Child currently on oral or IV antibiotics (washout period of 4 weeks allowable once antibiotics completed). Participants who require antibiotics after being enrolled in the study may continue on the study as usual.
* Immunodeficient disorders.
* Chronic disorder involving the gastrointestinal tract (e.g., inflammatory bowel disease, short gut syndrome, cystic fibrosis).
* Known hypersensitivity to components contained in study product.

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving treatment success | Between baseline and 12 weeks
  Clinically meaningful reduction (>= 8.7 points) in SCORAD index between baseline and 12 weeks without the use of rescue medication (systemic immunosuppression and/or biologic agents)

SECONDARY OUTCOMES:
Mean change in SCORAD index | From baseline to 12 weeks or time of starting rescue medication (whichever occurs earlier)
  Mean change from baseline to 12 weeks (or time of starting rescue medication, whichever occurs earlier) in Scoring Atopic Dermatitis (SCORAD) index
First use of rescue medication | From baseline to time of starting rescue medication (up to 12 weeks)
  Time from baseline to first use of rescue medication, up to 12 weeks
Mean change in RECAP | From baseline to 12 weeks or time of starting rescue medication (whichever occurs earlier)
  Mean change from baseline to 12 weeks (or time of starting rescue medication, whichever occurs earlier) in Recap of Atopic Eczema (RECAP) score. The RECAP score ranges from a minimum of 0 to a maximum of 28, with higher scores indicating worse outcomes.
Mean change in IDQOL | From baseline to 12 weeks or time of starting rescue medication (whichever occurs earlier)
  Mean change from baseline to 12 weeks (or time of starting rescue medication, whichever occurs earlier) in Infant Dermatitis Quality of Life (IDQOL) score. The IDQOL score ranges from a minimum of 0 to a maximum of 30, with higher scores indicating worse outcomes.
Mean change in EASI | From baseline to 12 weeks or time of starting rescue medication (whichever occurs earlier)
  Mean change from baseline to 12 weeks (or time of starting rescue medication, whichever occurs earlier) in Eczema Area and Severity Index (EASI) score. The EASI score ranges from a minimum of 0 to a maximum of 72, with higher scores indicating worse outcomes.
Mean change in IGA | From baseline to 12 weeks or time of starting rescue medication (whichever occurs earlier)
  Mean change from baseline to 12 weeks (or time of starting rescue medication, whichever occurs earlier) in Investigator Global Assessment for Atopic Dermatitis (IGA) score. The IGA score ranges from a minimum of 0 to a maximum of 4, with higher scores indicating worse outcomes.
Mean change in POEM | From baseline to 12 weeks or time of starting rescue medication (whichever occurs earlier)
  Mean change from baseline to 12 weeks (or time of starting rescue medication, whichever occurs earlier) in Patient-Oriented Eczema Measure (POEM) score. The POEM score ranges from a minimum of 0 to a maximum of 28, with higher scores indicating worse outcomes.
Use of topical corticosteroids | From baseline to 12 weeks
  Mean weight (in grams) of topical corticosteroids used by participants during the 12 weeks of the study.
Mean change in TOPICOP score | From baseline to 12 weeks or time of starting rescue medication (whichever occurs earlier)
  Mean change from baseline to 12 weeks in the Topical Corticosteroid Phobia (TOPICOP) score. The TOPICOP score ranges from a minimum of 0 to a maximum with 100, with higher scores indicating greater levels of phobia.
Mean change in gut microbiota | From baseline to 12 weeks or time of starting rescue medication (whichever occurs earlier)
  Mean change from baseline to 12 weeks (or time of starting rescue medication, whichever occurs earlier) in alpha diversity, beta diversity and short chain fatty avid levels measured from stool samples
Mean change in skin microbiota | From baseline to 12 weeks or time of starting rescue medication (whichever occurs earlier)
  Mean change from baseline to 12 weeks (or time of starting rescue medication, whichever occurs earlier) in alpha and beta diversity measured from skin swabs

CONTACTS AND LOCATIONS:
Overall Officials: Keith CY Ooi, Principal Investigator — University of New South Wales
Locations (1):
- Sydney Children's Hospital, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No